CLINICAL TRIAL: NCT05038202
Title: Study on the Efficacy and Safety of Bencycloquidium Bromide Nasal Spray Alone or in Combination With Mometasone Furoate Aqueous Nasal Spray in the Treatment of Moderate-severe Persistent Allergic Rhinitis
Brief Title: Study of Bencycloquidium Bromide Nasal Spray in the Treatment of Moderate-severe Persistent Allergic Rhinitis
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yingu Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YG-BLT-PMS001
Record Dates: First submitted 2021-08-23; First posted 2021-09-08 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Allergic Rhinitis
Keywords: allergic rhinitis; Bencycloquidium Bromide Nasal Spray
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Mometasone Furoate

STUDY DESIGN:
Intervention Model Description: 450 subjects with moderate-severe persistent allergic rhinitis will be enrolled in the trial and divided into three groups for different treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bencycloquidium Bromide (Experimental): Bencycloquidium Bromide Nasal Spray (90μg per spray)：1 spray on each nostril, 4times per day, continuous treatment for 4 weeks (28days).
  Interventions: Drug: Bencycloquidium Bromide Nasal Spray
- Mometasone Furoate Aqueous (Active Comparator): Mometasone Furoate Aqueous Nasal Spray (50μg per spray)：2 sprays on each nostril, 1 time per day, continuous treatment for 4 weeks (28days).
  Interventions: Drug: Mometasone Furoate Aqueous Nasal Spray
- Bencycloquidium Bromide with Mometasone Furoate Aqueous (Experimental): Bencycloquidium Bromide Nasal Spray in combination with Mometasone Furoate Aqueous Nasal Spray: For Bencycloquidium Bromide Nasal Spray(90μg per spray), 1 spray on each nostril, 4times per day. For Mometasone Furoate Aqueous Nasal Spray (50μg per spray), 2 sprays on each nostril, 1 time per day. If there is an overlap between the two drugs, use Bencycloquidium Bromide Nasal Spray first, and then mometasone furoate nasal spray should be used after an interval of more than 30 minutes.
  Interventions: Drug: Bencycloquidium Bromide Nasal Spray; Drug: Mometasone Furoate Aqueous Nasal Spray

INTERVENTIONS:
Drug: Bencycloquidium Bromide Nasal Spray — The content of this product is a colorless and clear liquid, press the sprayer, the liquid will be sprayed out in mist.
  This product is suitable for improving the symptoms of runny nose, nasal congestion, nasal itching and sneezing caused by allergic rhinitis.
  Other Names: BILITING
  Arms: Bencycloquidium Bromide; Bencycloquidium Bromide with Mometasone Furoate Aqueous
Drug: Mometasone Furoate Aqueous Nasal Spray — Mometasone furoate nasal spray is a quantitative hand-press spray device, and the content is a white to off-white suspension.
  This product is suitable for the treatment of seasonal or perennial rhinitis in adults, adolescents and children from 3 to 11 years old. For patients who have had moderate to severe seasonal allergic rhinitis symptoms, it is recommended to use this product 2-4 weeks before the start of the pollen season Preventive treatment.
  Other Names: NASONEX
  Arms: Bencycloquidium Bromide with Mometasone Furoate Aqueous; Mometasone Furoate Aqueous

SUMMARY:
450 subjects with moderate-severe persistent allergic rhinitis will be enrolled in the trial and divided into three groups for different treatments. Group A：Subjects with Bencycloquidium Bromide Nasal Spray, Group B：Subjects with Mometasone Furoate Aqueous Nasal Spray, Group C：Subjects with Bencycloquidium Bromide Nasal Spray in combination with Mometasone Furoate Aqueous Nasal Spray.The main purpose of the trial is to evaluate the efficacy of Bencycloquidium Bromide Nasal Spray alone or in combination with Mometasone Furoate Aqueous Nasal Spray in the treatment of moderate-severe persistent allergic rhinitis and rhinorrhea.

DETAILED DESCRIPTION:
The Secondary purpose is to evaluate the effectiveness of Bencycloquidium Bromide Nasal Spray alone or in combination with Mometasone Furoate Aqueous Nasal Spray in the treatment of moderate-severe persistent allergic rhinitis with nasal itching, nasal congestion, and sneezing. And evaluate the safety of Bencycloquidium Bromide Nasal Spray alone or in combination with Mometasone Furoate Aqueous Nasal Spray.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of allergic rhinitis meets the standards of "Guidelines for the Diagnosis and Treatment of Allergic Rhinitis" (2015, Tianjin);
* The previous or current symptom onset is ≥4d/week and ≥4 consecutive weeks; the symptoms are severe or serious (Total Nasal Symptom Scores≥6 points) with single symptom score of runny nose ≥2 points;
* Able to complete the symptom score as required;
* Subjects voluntarily participate in this study, and sign a written informed consent form. Use study drugs, complete evaluation and follow-up in accordance with the requirements of this study.

Exclusion Criteria:

* Those who are known to be allergic to the ingredients contained in test drugs.
* Used vasoconstrictors within 1 day; used topical or oral antihistamines within 3 days; used topical glucocorticoids and leukotriene receptor antagonists within 7 days; used oral glucocorticoid drugs within 30 days.
* Those who have been diagnosed as asthma or have asthma symptoms (wheezing, shortness of breath, chest tightness, coughing).
* Patients suffering from respiratory infections or abnormal nasal anatomy (such as nasal polyps, nasal septum deviation, etc.) one month before enrollment.
* Received immunotherapy and nasal surgery Within 6 months before enrollment.
* Patients with dry eye.
* Patients with glaucoma.
* Patients with enlarged prostate who have difficulty urinating.
* People with mental disorders or impaired consciousness.
* Pregnancy (patients report pregnancy), those who have a pregnancy plan within 6 months, and lactating women.
* Patients considered by the researcher to be unsuitable to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2021-06-16 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events | From the start of the enrollment to the end of the study, an average of 35days
  adverse clinical events that occur during drug treatment, which may not have a causal relationship with the drug.
Symptom scores of runny nose | immediately after the final intervention
  It is the symptom scores of runny nose, based on a 4-point method:
  0 points: asymptomatic;
  1. point: mild symptoms (symptoms are mild and easy to tolerate);
  2. points: moderate symptoms (significant symptoms, annoying, but tolerable);
  3. points: Severe symptoms (symptoms cannot be tolerated, affecting daily life and/or sleep).

SECONDARY OUTCOMES:
Visual Analogue Scale score of runny nose,nasal congestion, nasal itching, and sneezing | immediately after the final intervention
  Visual Analysis Scale (VAS, Visual Analysis Scale) score, from 0 to 10 points, the total symptoms of nasal congestion, nasal itching, and sneezing gradually increase; 0 of which is asymptomatic; 3 and below 3-the symptoms are mild and can be tolerated; 4 to 6 - the symptoms are severe but tolerable; 7 to 10 -symptoms are severe and unbearable, which affect appetite and sleep. The subjects calibrate it according to the intensity of the symptoms
Visual Analogue Scale score of total nasal symptoms | immediately after the final intervention
  24-hour retrospective review of the average change in the Visual Analogue Scale score of total nasal symptoms compared to the baseline. From 0 to 10 points, 0 of which is asymptomatic; 3 and below 3-the symptoms are mild and can be tolerated; 4 to 6 - the symptoms are severe but tolerable; 7 to 10 -symptoms are severe and unbearable, which affect appetite and sleep. The subjects calibrate it according to the intensity of the symptoms
Total Nasal Symptom Scores and Drug score | immediately after the final intervention
  Total nose symptom TNSS(Total Nasal Symptom Scores):
  It is the sum of 4 individual symptom scores of runny nose, nasal congestion, nasal itching and sneezing, totaling 12 points, and each symptom score is based on a 4-point method:
  0 points: asymptomatic;
  1. point: mild symptoms (symptoms are mild and easy to tolerate);
  2. points: moderate symptoms (significant symptoms, annoying, but tolerable);
  3. points: Severe symptoms (symptoms cannot be tolerated, affecting daily life and/or sleep).
  Drug score:
  0 points: No other drugs used to treat Allergic Rhinitis;
  1. point: Use oral antihistamines (Loratadine tablets designated in the trial, trade name: Claritin);
  2. points: use nasal hormones (not applicable for this trial);
  3. points: use oral hormones (not applicable for this trial).
The questionnaire of patient with global impression of change | immediately after the final intervention
  the subject's overall impression of symptoms change. From 0 to 4: 0 points: not evaluated;
  1. point: the symptoms are completely controlled or disappeared;
  2. points: Significant improvement in symptoms;
  3. points: the improvement of symptoms is not obvious;
  4. points: Symptoms are not improved or even worsened.
The questionnaire of Rhinoconjunctivitis Quality of Life | immediately after the final intervention
  the quality of sleep, symptoms of eyes, feelings of emotions due to the influence of nasal symptoms. From 0-6: 0-1 points: almost asymptomatic; 2-3 point: mild symptoms (symptoms are mild and easy to tolerate); 4-5 points: moderate symptoms (significant symptoms, annoying, but tolerable); 6 points: Severe symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Doctor, Principal Investigator — Beijing Tongren Hospital,CMU
Locations (6):
- China (6):
  - Beijing friendship hospital, CMU, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital,CMU, Beijing, Beijing Municipality
  - Beijing Tongren Hospital,CMU, Beijing, Beijing Municipality
  - The third affliation hospital of Sun YAT-SEN university, Guangzhou, Guangdong
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province hospital, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No